CLINICAL TRIAL: NCT06892171
Title: The Study of the Phenotype of Hereditary Xerocytosis
Acronym: EPIOX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Kremlin-Bicetre Hospital, Paris (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PI2023_843_0142
Record Dates: First submitted 2025-03-18; First posted 2025-03-24 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-03

CONDITIONS: Xerocytosis; Phenotype; Genotype
Keywords: xerocytosis; phenotype; genotype; PIEZO1; KCNN4 mutation
MeSH Terms: conditions — Xerocytosis, hereditary | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Biological: Blood sample — blood sample for genetic analysis

SUMMARY:
Hereditary xerocytosis is a dominant red blood cell membrane disorder characterized by an increased leakage of potassium from the interior to the exterior of the red blood cell membrane, leading to water loss, red cell dehydration, and chronic hemolysis. In 90% of cases, it is associated with heterozygous gain-of-function mutations in PIEZO1, a gene that encodes a mechanotransducer responsible for converting mechanical stimuli into biological signals. The remaining 10% of cases are linked to mutations in the GARDOS channel gene.

ELIGIBILITY:
Inclusion Criteria:

* Any patient diagnosed with hereditary xerocytosis according to the 2021 PNDS guidelines
* Covered by a social security plan
* Signature of the consent form for study participation by the patient, or for minors, by the parent(s)/legal representative(s).

Exclusion Criteria:

* patients with other hemolysis reason

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
identification of PIEZO1 mutations | 36 months
identification of KCNN4 mutations | 36 months
correlation between the identified PIEZO1 mutations and Hemoglobin levels | 36 months
correlation between the identified KCNN4 mutations and Hemoglobin levels | 36 months
correlation between the identified PIEZO1 mutations and reticulocytes levels | 36 months
correlation between the identified KCNN4 mutations and reticulocytes levels | 36 months
correlation between the identified PIEZO1 mutations and Ferritin levels | 36 months
correlation between the identified KCNN4 mutations and Ferritin levels | 36 months
correlation between the identified PIEZO1 mutations and MRI quantification of intrahepatic iron | 36 months
correlation between the identified KCNN4 mutations and MRI quantification of intrahepatic iron | 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No